CLINICAL TRIAL: NCT05519566
Title: The Diagnostic Accuracy of Pulsed Fluoroscopy Retrograde Urethrogram Vs the Traditional Retrograde Urethrogram In Diagnosing Urethral Stricture: A Randomized Prospective Comparative Study
Brief Title: The Accuracy of Pulsed Fluoroscopy Retrograde Urethrogram Vs the Traditional Retrograde Urethrogram In Diagnosing Urethral Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Ontario School of Medicine (Other)
Responsible Party: Principal Investigator, Walid Shahrour, Associate professor, Northern Ontario School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021515
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Urethral Stricture
Keywords: Diagnosing Urethral Stricture; Pulsed Fluoroscopy Retrograde Urethrogram; Traditional Retrograde Urethrogram
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Fluoroscopy Retrograde Urethrogram (Experimental)
  Interventions: Diagnostic Test: Retrograde Urethrogram
- Traditional Retrograde Urethrogram (Active Comparator)
  Interventions: Diagnostic Test: Retrograde Urethrogram

INTERVENTIONS:
Diagnostic Test: Retrograde Urethrogram — Fluoroscopy Retrograde Urethrogram Vs the Traditional Retrograde Urethrogram

SUMMARY:
This study is designed as a prospective comparative randomized clinical study to determine the diagnostic accuracy (sensitivity, specificity, positive predictive value, and negative predictive value) of pulsed fluoroscopy retrograde urethrogram for urethral stricture disease. The target population includes patients scheduled for retrograde urethrogram either new referral or follow up at Thunder Bay Regional Health Sciences Centre (TBRHSC) for treatment of urethral stricture who meet the specific eligibility criteria. The overall number of participants targeted will be 46. Upon presentation to the urology clinic or ambulatory care unit, the treating urologist/investigator will notify the patient of an opportunity to participate in the study. If the patient is interested, a research team member who is not directly involved in the patient care will be invited to discuss the study to the potential participant.

The study team member will obtain a full-informed consent form the potential participant.

Following informed consent, participants will be screened to ensure they meet the specific eligibility requirements of this study, through consultation with their medical records and the treating urologist. Randomization will be conducted in a 1:1 allocation ratio to either treatment arm: (1) the Pulsed fluoroscopy retrograde urethrogram, or (2) the Traditional retrograde urethrogram.

Using an Excel sheet, the RAND function will give a random code. The random code is a figure ranging from 0.00000000 to 0.9999999999. A 0.5 cut-off code will be used, below which we will use the small blocks of 4 cells (4 rows of excel) and above which we will use the large blocks of 8 cells (8 rows of excel). Participants will undergo procedures according to the order of randomization Participants will undergo either Pulsed fluoroscopy retrograde urethrogram or Traditional retrograde urethrogram, depending on the treatment arm they are randomized to. Clinical data such as stricture location, stricture length and possible adverse effects will be recorded. According to the urologist decision based on data obtained during RUG, participant will be scheduled for urethroplasty or cystoscopy. All participants will undergo these procedures according to standard care procedures at TBRHSC.

Data collection at baseline will include demographics, and relevant medical history. All retrograde urethrogram data including the type of urethrogram, the urethrogram date, fluoroscopy time, cumulative radiation dose, stricture location, stricture length and intraprocedural complications.

Furthermore, we will record intraoperative data such as operative date, stricture location and stricture length. De-identified research files will be maintained in a secure office of a research team member during the conduct of the study. De-identified research data will be input into an electronic database that is password protected and maintained on research team member's computers or encrypted USB devices. An enrolment log, linking Participant ID to identifiable information will be maintained in hard copy in a locked office, or electronically as a password-protected document on the TBRHSC network.

Only delegated research team members and the Principal Investigator will have access to research and patient data.

Upon study closure, research records will be kept in secure storage in a research team member's office for a period of 5 years. Following this, the files will be securely shredded, and any electronic documents permanently deleted.

Data will be analyzed using the commercially available SPSS software version 26 (SPSS Inc., Chicago, IL, USA). For both techniques, data obtained during baseline and postoperative urethrograms will be compared in terms of stricture location, stricture length, fluoroscopy time, cumulative radiation dose and the occurrence of intraprocedural complications. Categorical data will be compared using Chi-squared or Fisher test. Continuous data will be analyzed using the T test or Mann-Whitney U test

Data obtained during urethroplasty will set as a standard of comparison to determine sensitivity, specificity, positive predictive value and negative predictive value of pulsed fluoroscopy and traditional urethrograms. For each comparison, 2 × 2 contingency tables were used to present the results and calculate the diagnostic accuracy estimates with 95% confidence intervals Data analysis will be done blindly regarding the type of performed procedure. One procedure will be coded as "1" and the other will "2". Categorical variables will be presented using number and percentage, and continuous variables will be presented using median and ranges. Two-tailed p-values of less than 0.05 will be set for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Males over 18 years of age at the time of enrollment
* Referred to urology for a suspected diagnosis of stricture urethra.
* Ability to get written informed consent to participate
* Ability to comply with study procedures

Exclusion Criteria:

* Co-existing urethral fistula, or requiring fluoroscopic guided manipulation
* Active urinary tract infection not yet appropriately treated
* Pre-existing conditions, which, in the opinion of the investigator, interfere with the conduct of the study
* Lack of capacity to provide free and informed written consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 46 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of pulsed fluoroscopy retrograde urethrogram | Intra-procedure (during the urethroplasty)
  Sensitivity, specificity, positive predictive value, and negative predictive value of pulsed fluoroscopy retrograde urethrogram
diagnostic accuracy of pulsed traditional retrograde urethrogram | Intra-procedure (during the urethroplasty)
  Sensitivity, specificity, positive predictive value, and negative predictive value of pulsed traditional retrograde urethrogram

SECONDARY OUTCOMES:
Intraprocedural adverse events | Intra-procedure (during the urethroplasty)
  Any adverse events (e.g., extravasation of contrast)

CONTACTS AND LOCATIONS:
Locations (1):
- Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario, Canada